CLINICAL TRIAL: NCT01172418
Title: Randomized Trial of 2 Antibody Induction Steroid Avoidance Protocols Accompanied by Maintenance Therapy With Prograf® and Myfortic®
Brief Title: Randomized Trial of 2 Antibody Induction Steroid Avoidance Protocols
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, George W. Burke, Chief, Kidney and Kidney-Pancreas Transplantation, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #20057672
Record Dates: First submitted 2010-06-10; First posted 2010-07-29 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Transplant; Failure, Kidney
Keywords: adult; primary kidney transplant recipient
MeSH Terms: interventions — Alemtuzumab; Daclizumab; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymoglobulin and Daclizumab (Active Comparator): Group I: Our standard steroid avoidance protocol, i.e., 3 daily doses of 1 mg/kg of Thymoglobulin®, the first to be infused at surgery, accompanied by 2 doses of anti-CD25 humanized monoclonal antibody, the first also to be given at surgery, and the second 2 weeks later. (controls)
  Interventions: Drug: Daclizumab; Drug: Thymoglobulin
- Thymoglobulin and Alemtuzumab (Experimental): Group II: A new steroid avoidance protocol in which 1 dose of 1 mg/kg of Thymoglobulin® is to be infused at surgery followed by 1 dose of alemtuzumab (Campath-1H) at 0.3 mg/kg within 24 hours. No further antibody therapy will be used.
  Interventions: Drug: Alemtuzumab; Drug: Thymoglobulin

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab used as part of combined Induction.
  Other Names: Campath-1H (Alemtuzumab)
  Arms: Thymoglobulin and Alemtuzumab
Drug: Daclizumab — Daclizumab used as part of combined induction.
  Other Names: Zenapax (Daclizumab)
  Arms: Thymoglobulin and Daclizumab
Drug: Thymoglobulin — Thymoglobulin used as part of combined induction.
  Other Names: rATG (rabbit antithymocyte globulin)

SUMMARY:
The purpose of the present study is to determine which antibody induction regimen will result in a safer and more effective method to use with steroid avoidance in renal transplant recipients. Patients receiving either first cadaveric or non-HLA identical living donor kidney transplants will be preoperatively randomized into 2 groups.

DETAILED DESCRIPTION:
Antibody Induction:

Group I: Our standard steroid avoidance protocol, i.e., 3 daily doses of 1 mg/kg of Thymoglobulin®, the first to be infused at surgery, accompanied by 2 doses of anti-CD25 humanized monoclonal antibody, the first also to be given at surgery, and the second 2 weeks later. (controls) Group II: A new steroid avoidance protocol in which 1 dose of 1 mg/kg of Thymoglobulin® is to be infused at surgery followed by 1 dose of alemtuzumab (Campath-1H) at 0.3 mg/kg within 24 hours. No further antibody therapy will be used.

In both groups, Prograf® maintenance therapy will be rapidly initiated (vide-infra) with a targeting dosage to 12 hour trough levels of 4 to 8 ng/ml.

In Group I, maintenance dosing Myfortic® will be targeted to 720 mg twice daily. In Group II, maintenance doses of Myfortic® will be targeted to 360 mg twice daily.

Steroids are to be given equivalently in both groups only during the first week postoperatively. The regimen consists of 500 mg/day of Solumedrol intravenously for 3 postoperative days followed by daily oral methylprednisolone or IV Solumedrol at 1 mg/kg per day, decreasing to 0.5 mg/kg per day during the remainder of the week primarily to avoid hypersensitivity reactions to the induction antibodies. No further steroid use is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been fully informed and has signed a dated IRB approval informed consent form and is willing to follow study procedures for the extent of the study (12 months). Parent or legal guardian must provide written consent for patients <18 years of age.
2. Age 18-70 years
3. Weight > 40 kg
4. Primary renal allograft: living or deceased donor
5. Negative standard crossmatch for T cells. All deceased donor-recipient pairs matched for a minimum of 1 HLA DR antigen. (Standard at our center.)
6. Women of childbearing potential will be required to have a negative qualitative serum pregnancy test and agree to use an adequate method of contraception for the study duration.
7. Males and females are to be studied equivalently as they become available for transplantation using these criteria.

   -

Exclusion Criteria:

* 1. Patient has previously received or is receiving an organ transplant other than a kidney.

  2. Patient is receiving an ABO incompatible donor kidney. 3. Recipient or donor is seropositive for human immunodeficiency (HIV), Hepatitis C viruses, or Hepatitis B virus antigenemia.

  4. Patient has a current malignancy or a history of malignancy (within the past 5 years), except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully, or carcinoma in situ of the cervix that has been treated successfully.

  5. Patients with significant liver disease, defined as having during the past 28 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of the normal range of this center.

  6. Patient has uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or an active peptic ulcer or any other unstable medical condition that could interfere with study objectives.

  7. Patient is currently participating in another clinical trial of an investigational drug in the 30 days prior to transplant.

  8. Patient will be receiving any immunosuppressive agent other than those prescribed in the study.

  9. Patient is unable to take medications orally or via nasogastric tube by the morning of the second day following completion of the transplant procedure (i.e., skin closure).

  10. Patient is receiving or may require warfarin, fluvastatin, or herbal supplements during the study.

  11. Concurrent use of astemizole, pimozide, cisapride, terfenadine, or ketoconazole.

  12. Patient has a known hypersensitivity to tacrolimus, Thymoglobulin®, IL-2 receptor inhibitor monoclonal antibodies, alemtuzumab, sirolimus, MMF, Myfortic®, or corticosteroids.

  13. Patient is pregnant or lactating. 14. Patients with a screening/baseline (or within 96 hours of transplant) total white blood cell count <4000/mm3; platelet count <100,000/mm3; fasting triglycerides >400 mg/dl (>4.6 mmol/L); fasting total cholesterol >300 mg/dl (>7.8 mmol/L); fasting HDL-cholesterol <30 mg/dl; fasting LDL-cholesterol >200 mg/dl.

  15. Patient is unlikely to comply with the visits scheduled in the protocol. 16. Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.

  17. If tacrolimus cannot be instituted for longer than 5 days postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

REFERENCES:
- [Result] Ciancio G, Gaynor JJ, Sageshima J, Guerra G, Zarak A, Roth D, Brown R, Kupin W, Chen L, Hanson L, Tueros L, Ruiz P, Livingstone AS, Burke GW 3rd. Randomized trial of dual antibody induction therapy with steroid avoidance in renal transplantation. Transplantation. 2011 Dec 27;92(12):1348-57. doi: 10.1097/TP.0b013e3182384b21. PMID 22027927

RESULTS

PARTICIPANT FLOW:
Groups:
- Thymoglobulin and Daclizumab: Group I: Our standard steroid avoidance protocol, i.e., 3 daily doses of 1 mg/kg of Thymoglobulin®, the first to be infused at surgery, accompanied by 2 doses of anti-CD25 humanized monoclonal antibody, the first also to be given at surgery, and the second 2 weeks later. (controls)
  Daclizumab: used in combination with Thymoglobulin as combined induction
- Thymoglobulin and Alemtuzumab: Group II: A new steroid avoidance protocol in which 1 dose of 1 mg/kg of Thymoglobulin® is to be infused at surgery followed by 1 dose of alemtuzumab (Campath-1H) at 0.3 mg/kg within 24 hours. No further antibody therapy will be used.
  Alemtuzumab: used in conjunction with Thymoglobulin as combined Induction.
Period: Overall Study
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Started | 100 | 100
Completed | 100 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis performed on all 200 patients in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: participants] | 49.9 (12) | 49.4 (13) | 49.65 (12.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 91 | 87 | 178
  >=65 years | 9 | 13 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 72 | 76 | 148
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Rejection at One Year Post-transplant
Time Frame: at one year post-transplant
Measure: Number; unit: percentage of patients having BPAR
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Number analyzed (Participants) | 100 | 100
percentage of patients having BPAR | 14 | 13

2. Secondary Outcome: Graft Survival
Time Frame: at 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: actuarial percentage of participants
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Number analyzed (Participants) | 100 | 100
actuarial percentage of participants | 92.9 [87.9 to 98.0] | 92.0 [86.7 to 97.3]
Statistical Analysis 1: Comparison: Thymoglobulin and Daclizumab vs Thymoglobulin and Alemtuzumab; Test type: Superiority; p = 0.78, Log Rank

3. Secondary Outcome: Graft Survival
Time Frame: at 3 years post-transplant
Measure: Number (95% Confidence Interval); unit: actuarial percentage of participants
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Number analyzed (Participants) | 100 | 100
actuarial percentage of participants | 90.9 [85.2 to 96.5] | 86.9 [80.2 to 93.5]
Statistical Analysis 1: Comparison: Thymoglobulin and Daclizumab vs Thymoglobulin and Alemtuzumab; Test type: Superiority; p = 0.37, Log Rank

4. Secondary Outcome: Patient Survival
Time Frame: at 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: actuarial percentage of participants
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Number analyzed (Participants) | 100 | 100
actuarial percentage of participants | 96.9 [93.5 to 100.4] | 97 [93.6 to 100.4]
Statistical Analysis 1: Comparison: Thymoglobulin and Daclizumab vs Thymoglobulin and Alemtuzumab; Test type: Superiority; p = 0.99, Log Rank

5. Secondary Outcome: Patient Survival
Time Frame: at 3 years post-transplant
Measure: Number (95% Confidence Interval); unit: actuarial percentage of participants
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Number analyzed (Participants) | 100 | 100
actuarial percentage of participants | 95.9 [91.9 to 99.8] | 91.8 [86.4 to 97.3]
Statistical Analysis 1: Comparison: Thymoglobulin and Daclizumab vs Thymoglobulin and Alemtuzumab; Test type: Superiority; p = 0.25, Log Rank

ADVERSE EVENTS:
Description: Total Numbers at Risk for Serious Adverse Events (100+100=200) and Other Adverse Events (75+70=145) were inconsistent, because in order to determine how many study participants developed NODAT (new onset diabetes after transplant), study participants having pre-transplant diabetes (25 in Groups I, and 30 in Group II) were excluded.
Arm/Group | Thymoglobulin and Daclizumab | Thymoglobulin and Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 29/100 | 25/100
Other Adverse Events (participants affected / at risk) | 8/75 | 8/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoglobulin and Daclizumab (N=100) | Thymoglobulin and Alemtuzumab (N=100)
Patients who developed an infection that required hospitalization (Infections and infestations) | 29 | 25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoglobulin and Daclizumab (N=75) | Thymoglobulin and Alemtuzumab (N=70)
occurrence of NODAT in patients without pretransplant diabetes (Endocrine disorders) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No